CLINICAL TRIAL: NCT03870490
Title: An Open-Label Trial to Assess the Safety and Pharmacokinetics of VNRX-5133 in the Epithelial Lining Fluid of Healthy Adult Subjects
Brief Title: Safety and Pharmacokinetics of VNRX-5133 in the Epithelial Lining Fluid of Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VNRX-5133-106; 272201300019C-17-0-3 (NIH); 18-0001 (Other: DMID)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — taniborbactam; Cefepime

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): VNRX-5133 + cefepime
  Interventions: Drug: VNRX-5133 + cefepime

INTERVENTIONS:
Drug: VNRX-5133 + cefepime — IV infusion (3 doses)

SUMMARY:
This is a single-center, open-label study to assess safety and pharmacokinetics of VNRX-5133 and cefepime in the epithelial lining fluid in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the trial, give written informed consent, and comply with the trial restrictions
* Gender: male or female with a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at Screening and Day -1; females may be of childbearing potential or of nonchildbearing potential
* Age: ≥18 years at Screening
* Weight: ≥50 kg
* Body mass index (BMI): ≥18 kg/m2 and <30 kg/m2
* Normal blood pressure (BP), defined as a systolic value ≥90 mm Hg and ≤140 mm Hg and a diastolic value <90 mm Hg (Screening and Day -1)
* All values for hematology and clinical chemistry tests of blood and urine are either within normal limits of laboratory reporting range (WNL) or defined as permitted exceptions
* Ability and willingness to abstain from alcohol, from 48 hours (2 days) prior to admission to the Clinical Research Center (CRC) until discharge from the CRC
* Males who are not surgically sterilized and females of childbearing potential must agree to use highly effective methods of contraception during this trial and for 90 days after the last dose of study drug
* All over-the-counter (OTC) medications, health supplements, and herbal remedies (eg, St. John's Wort extract) must have been stopped at least 14 days prior to admission to the CRC
* Suitable veins for cannulation/multiple venipunctures as assessed by the Investigator at Screening

Exclusion Criteria:

* Employee of the Contract Research Organization (CRO), CRC, or the Sponsor
* Female who is pregnant, lactating, or at risk of becoming pregnant during this trial or within 90 days after the last dose of study drug
* Male with a female partner who is pregnant or lactating during this trial or planning to attempt to become pregnant during this trial or within 90 days after the last dose of study drug
* Use of any investigational drug or device within 30 days prior to Screening (90 days for an injectable biological agent)
* Presence of a congenital or acquired immunodeficiency syndrome
* Any evidence or history of clinically significant medical abnormalities on PE or laboratory assessment
* Clinically significant ECG abnormality
* Sitting systolic BP >140 mm Hg or diastolic BP >90 mm Hg on a single measurement following at least 5 minutes of rest at Screening
* History of drug allergy of a severity that required urgent medical treatment such as treatment with epinephrine in an Emergency Department
* History of any hypersensitivity reaction following administration of a cephalosporin, penicillin, or other β-lactam antibacterial drug or any component of VNRX-5133 for injection formulation
* History of hypersensitivity to lidocaine, midazolam, fentanyl, or other topical anesthetics/opioids in similar classes to these agents
* Use of prescription or nonprescription drugs, vitamins, or dietary supplements within 14 days prior to the first dose of study drug
* History of donation of >450 mL of blood within 60 days prior to first dose of study drug or planned donation before 30 days has elapsed since final dose of study drug
* Plasma or platelet donation within 7 days of first dose of study drug or planned donation during this trial
* Current suspected drug or alcohol abuse as specified in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision criteria
* Recent history of alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 standard drink=5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months before Screening
* Use of tobacco- or nicotine-containing products from Screening through Check Out

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) in Epithelial Lining Fluid (ELF) | Day 2
  Steady-state plasma PK and disposition of cefepime/VNRX-5133 in the ELF
Safety as measured by the number of subjects with adverse events | Days 1-7
  Number of Subjects with AEs (Assessed via patient report, physical exam, ECGs, vital signs, laboratory investigations, and use of concomitant medications for the treatment of AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No